CLINICAL TRIAL: NCT01589250
Title: Risk Scoring Systems in Upper GI-haemorrhage
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stig Borbjerg Laursen, MD, Odense University Hospital
Other Study IDs: SBL-03
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Upper Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Use of risk scoring systems in the assessment of patients presenting with upper gastrointestinal haemorrhage is increasing. Comparative studies have intended to identify the system of choice, but the majority of these are characterized by retrospective designs, small sample sizes, low rate of severe bleeding, or low mortality. The main aim of this study was to identify the optimal scoring system.

ELIGIBILITY:
Inclusion Criteria:

One of the following:

* Haematemesis
* Melaena
* Coffee-ground vomit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data were collected from consecutive patients admitted with UGIH at Odense University Hospital between August 2009 and August 2011. UGIH was defined as history of haematemesis, coffee-ground vomit, or melaena.
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Need for hospital-based intervention | 1 month
  Need of hospital-based intervention was defined as treatment with blood transfusion, endoscopic therapy, transcatheter arterial embolization (TAE), surgery, or identification of cancer at upper endoscopy.

SECONDARY OUTCOMES:
Identification of low-risk patients | 1 month
  Low-risk patients were defined as patients who did not need hospital-based intervention, and survived more than 30 days from day of admission. Low-risk patients were considered as suitable for early discharge and potential outpatient management.
Rebleeding | 1 month
  Rebleeding was defined as presence of hematemesis, blood per nasogastric tube, or melaena associated with a decline in B-hemoglobin of at least 1mmol/l (not explained by hemodilution) or decline in systolic arterial pressure of at least 20mmHg after the initial bleeding had stopped.
30 day mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Laursen SB, Hansen JM, Schaffalitzky de Muckadell OB. The Glasgow Blatchford score is the most accurate assessment of patients with upper gastrointestinal hemorrhage. Clin Gastroenterol Hepatol. 2012 Oct;10(10):1130-1135.e1. doi: 10.1016/j.cgh.2012.06.022. Epub 2012 Jul 16. PMID 22801061